CLINICAL TRIAL: NCT06605183
Title: 10,000 STEP CLUB: Community Walking Program to Decrease Sedentary Behavior, Fear of Falling Avoidance Behavior, Loneliness, and Social Isolation in Parkinson's Disease
Brief Title: 10,000 Step Club: Community Walking Program for People with Parkinson's Disease
Acronym: (10KSC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Merrill Landers, Primary investigator, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLVPT 10KSC
Record Dates: First submitted 2024-09-12; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
Keywords: Exercise; Nordic walking; physical activity; social isolation; loneliness; fear of falling; walking
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One hour per week of community walking for 6 months (Other): Participants will participate in one, 60-minute group walk using Nordic poles at a local community park. Participants will be assessed before and after the 6-month program.
  Interventions: Behavioral: Community walking program using Nordic walking poles

INTERVENTIONS:
Behavioral: Community walking program using Nordic walking poles — This is a group, community walking program at local parks using Nordic walking poles. Participants will be encouraged to walk briskly but safely for 60 minutes one time per week with the ultimate goal of using this community walking program to build up their step count to 10,000 steps per day. We do not anticipate that the weekly walk will get them to 10,000 steps but we will use that as a weekly event to drive behavioral change throughout the week.

SUMMARY:
The 10,000 Step Club (10KSTC) is a 6-month community walking program for people with Parkinson's disease (PwP) and their caregivers in Las Vegas, Nevada (LV). This program will consist of several weekly, organized walking groups in local parks throughout the LV Valley. Participants in the program will use Nordic walking poles during the walks. Each walking group will meet once per week at a local park and will be supervised by walking group leaders from the University of Nevada, Las Vegas. There will be three walking programs throughout the Las Vegas valley. Participants will be given a step watch to wear step counts will be tracked in real-time. The program is designed to get PwP out of their homes, cultivate a culture of connection with others with Parkinson's disease (PD), and to be collectively accountable for a common goal toward 10,000 steps per day.

DETAILED DESCRIPTION:
The 10,000 Step Club (10KSC) is a 6-month community walking program conducted at various local parks in Las Vegas (LV), Nevada for people with Parkinson's disease (PD). There will be three walking groups and each group will meet at a local park once weekly for a 60-minute walk. These walking groups will be led by UNLV physical therapy students who will organize, coordinate, and manage the different walking groups. Participants will be encouraged to attend at least one walking group per week in their area but will be permitted to participate at the other walking groups on different days if they desire to get in a second or third walk that week. Participants in the program will use Nordic walking poles to promote stability and upright posture, and to encourage full body movement and arm use.

There will be three different walking groups throughout Las Vegas in areas with few PD exercise programs and higher proportions of people with Parkinson's disease in lower socioeconomic regions and historically underserved areas. The 10KSC program will be offered in both English and Spanish. Participants will be given a step watch to wear over the 6 months of the program and will be encouraged to build up their physical activity to eventually average 10,000 steps per day. The watches will be used to track step counts in real-time and there will be an incentive program to motivate participants and recognize achievements related to program goals. The program is designed to get people with Parkinson's disease out of their homes, cultivate a culture of connection with others with Parkinson's disease to decrease social isolation and loneliness, and to be collectively accountable for a common goal toward more physical activity. The 10KSC will be evaluated for effectiveness, feasibility, and safety. The program will target recruitment of 60 participants with Parkinson's disease. Participation will be free of charge and care partners will be encouraged to participate as well. The program inclusion criteria will be "pragmatic" which means that there will be few exclusion criteria and the only inclusion criterion will be a diagnosis of Parkinson's disease by a neurologist.

ELIGIBILITY:
Inclusion Criteria:

* 30-85 years old
* Neurologist-diagnosed Parkinson's disease
* Able to walk independently with or without a walking aid (e.g., cane, walker)
* Willing to participate in a 6-month study

Exclusion Criteria:

* Health diagnosis that would limit exercise participation (e.g., heart problems, uncontrolled blood pressure, exercise-induced asthma).
* Dementia. This will be determined by completing the Montreal Cognitive Assessment
* Participants with poor walking ability (determined using the Timed Up and Go Test during initial testing).

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Daily step count average | From enrollment to the end of the 6-month community walking program.
  Daily step count average over one week as determined using a step watch and using real-time data acquisition software.
Fear of Falling Avoidance Behavior | From enrollment to the end of the 6-month community walking program.
  This will be assessed using the modified Fear of Falling Avoidance Behavior Questionnaire which is a self-report scale ranging from 0 to 56 with higher scores suggestive of more fear of falling avoidance behavior.
Social isolation | From enrollment to the end of the 6-month community walking program.
  Patient-Reported Outcomes Measurement Information System (PROMIS) v2.0 - Social Isolation - Short Form 8a. This is a self-report questionnaire ranging from 8 to 40 with higher scores suggestive of more social isolation.
Loneliness | From enrollment to the end of the 6-month community walking program.
  Patient-Reported Outcomes Measurement Information System (PROMIS) v2.0 - Loneliness - Fixed Form. This is a self-report questionnaire with scores ranging from 5 to 25 with higher scores suggestive of more loneliness.
Self-efficacy | From enrollment to the end of the 6-month community walking program.
  Patient-Reported Outcomes Measurement Information System (PROMIS) v1.0 - Self-Efficacy for Chronic Conditions - Managing Emotions - Short Form 8a. This is a self-report questionnaire with scores ranging from 8 to 40 with higher scores suggestive of more self-efficacy.

SECONDARY OUTCOMES:
Program goals - feasibility | Through the completion of the study, an average of 6-months.
  Number of participants that started and completed the 6-month program (75% of enrollees will complete the full, 6-month program).
  Percent week-to-week attendance of the schedule walking days (75% of the participants will have attended at least 75% of the weekly walks (one required per week)).
  Percent of participants who wear the step watch more than 20 hours per day (75% of the participants will be compliant with wearing the step watch for at least 20 hours per day).
  Percentage of participants who felt the program was beneficial and worthwhile. (75% of the participants who completed the program will agree or strongly agree that the program was beneficial and worthwhile).
Program goals - safety | Through the completion of the study, an average of 6-months.
  Number of falls and other injuries sustained during the weekly walks.
  1. 75% of the participants will have not sustained a fall or injury during participation in the weekly walks.
  2. 75% of the participants will not have sustained a musculoskeletal injury requiring medical attention related to the program.
Enrollment goals - diversity | Through the completion of the study, an average of 6-months.
  Participation of Black/African American PwP. 1. Recruitment will be deemed a success if at least 8 participants who identify as Black/African American are recruited and retained. This number is based on the percent of people in LV who identify as Black/African American (12.9%).
  Participation of Hispanic/Latino/Latina PwP.
  1. Recruitment will be deemed a success if at least 20 participants who identify as Hispanic/Latino/Latina are recruited and retained. This number is based on the percent of people in LV who identify as Hispanic/Latino/Latina (33.3%).

CONTACTS AND LOCATIONS:
Locations (1):
- Gait and Balance Laboratory, 217 Bigelow Health Sciences Building, UNLV, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided